CLINICAL TRIAL: NCT07380659
Title: Safety and Efficacy of Allogeneic Immunosuppressive CAR-DC Targeting FAP in the Treatment of Acute Myocardial Infarction With Cardiogenic Shock
Brief Title: Safety and Efficacy of FAP iCDC in Acute Myocardial Infarction With Cardiogenic Shock
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YAN2025-1716
Record Dates: First submitted 2026-01-05; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cardiogenic Shock; Cardiogenic Shock Post Myocardial Infarction; STEMI - ST Elevation Myocardial Infarction
Keywords: acute myocardial infarction with cardiogenic shock
MeSH Terms: conditions — Shock, Cardiogenic; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Administration of allogeneic FAP iCDC (Experimental): Administration of FAP immunosuppressive CAR-DC cell therapy in AMI CS. Patients are planned to be enrolled in the dose-escalation trial (1×10^5/kg、4×10^5/kg、and 8×10^5/kg) .The first dose group (4×10⁵/kg) initially enrolls 3 subjects to observe Dose-Limiting Toxicity (DLT) responses.
  1. If no DLT occurs and all 3 subjects demonstrate efficacy after 6 months of treatment, and this dose is determined as the safe and effective dose.
  2. If 1 subject experiences DLT, 3 additional subjects are enrolled. ·If 1/6 subjects develops DLT, and efficacy is not fully achieved in all 6 subjects, escalate to the next dose group (8×10^5/kg). ·If ≥2/6 subjects develop DLT, de-escalate to the previous dose group (1×10^5/kg).
  3. After identifying a safe and effective dose, enrollment will be expanded at this dose to bring the total sample size to 8-10 subjects, to further evaluate safety and efficacy.
  Interventions: Biological: FAP allogeneic immunosuppressive CAR-DC
- Standard therapy (No Intervention): Patients in the control group do not receive cellular therapy intervention.

INTERVENTIONS:
Biological: FAP allogeneic immunosuppressive CAR-DC — Each subject receive FAP immunosuppressive CAR-DC by intravenous infusion at the first day of shock.
  Arms: Administration of allogeneic FAP iCDC

SUMMARY:
To study the safety and efficacy of fibroblast activation protein (FAP)-targeted allogeneic immunosuppressive chimeric antigen receptor-dendritic cell (CAR-DC) in the treatment of acute myocardial infarction with cardiogenic shock and provide a new method for the treatment of acute myocardial infarction with cardiogenic shock.

DETAILED DESCRIPTION:
Background: Cardiogenic shock following acute myocardial infarction (AMI) remains a major unresolved clinical challenge. Despite advances in urgent revascularization and mechanical circulatory support, short-term mortality remains unacceptably high, approaching 40% within 30 days. Few evidence-based therapies have demonstrated a meaningful survival benefit, highlighting the urgent need for novel, mechanism-driven interventions. Growing clinical and experimental evidence indicates that a dysregulated systemic inflammatory response-manifested by hyperthermia, leukocytosis, and elevated proinflammatory mediators-plays a central role in the pathophysiology and progression of cardiogenic shock. Excessive inflammation exacerbates myocardial dysfunction, promotes multiorgan injury, and impairs recovery, suggesting that targeted immunomodulation may represent a complementary therapeutic strategy in this high-risk population. Dendritic cells (DCs), as professional antigen-presenting cells, occupy a pivotal position at the interface of innate and adaptive immunity and are uniquely suited to orchestrate context-dependent immune responses. In particular, tolerogenic DCs exert potent immunosuppressive effects through regulatory cytokine production, expression of co-inhibitory ligands, antigen-specific suppression of effector T cells, and induction of regulatory T cells. Collectively, these properties render DCs an attractive yet underexplored cellular platform for resolving excessive inflammation and promoting tissue repair in cardiogenic shock with AMI.

Purpose: In this prospective clinical study, the investigators engineered a stable, immunosuppressive, and fibrotic lesion-targeted DC therapy, termed immunosuppressive DCs (iCDC). This study was designed to evaluate the safety and preliminary efficacy of allogeneic fibroblast activation protein (FAP)-targeted iCDC therapy in patients with AMI complicated by cardiogenic shock.

Study design: This single-center, prospective, concurrent non-randomized controlled clinical trial enrolls patients aged 18-80 years presenting with acute myocardial infarction complicated by cardiogenic shock. Eligible patients are treated with allogeneic FAP-targeted immunosuppressive iCDC therapy.

Outcome measure: The primary outcome is the safety of FAP-targeted immunosuppressive iCDC therapy in patients with AMI complicated by cardiogenic shock. Secondary outcomes include 30-day all-cause mortality; hemodynamic parameters following iCDC therapy (systolic blood pressure, diastolic blood pressure, mean arterial pressure, and heart rate); time to hemodynamic stabilization; dose and duration of vasopressor and inotropic support; arterial lactate levels; changes in biomarkers (BNP, CRP, creatinine, ALT, AST, and inflammatory mediators); need for and duration of mechanical ventilation; need for and duration of left ventricular assist device implantation; intensive care unit and total hospital length of stay; left ventricular ejection fraction assessed by echocardiography; SAPS II score; SCAI shock classification; heart failure symptom burden assessed by NYHA functional class and the Kansas City Cardiomyopathy Questionnaire; incidence of major adverse cardiovascular events (MACE), including cardiac death and heart failure hospitalization; and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria（patients）:

* Age ≥ 18 years and < 80 years.
* Acute ST-segment elevation myocardial infarction (STEMI) complicated by cardiogenic shock, meeting all the following conditions:

  1. Post-emergent revascularization (PCI or CABG)
  2. Systolic blood pressure < 90 mmHg for >30 minutes, or requiring catecholamine support to maintain systolic blood pressure >90 mmHg
  3. Signs of impaired organ perfusion, meeting at least one of the following criteria:

     1. Altered mental status
     2. Cold, clammy skin and extremities
     3. Oliguria, with urine output <30 mL/h
     4. Arterial lactate level >2 mmol/L
* The patient or their legally authorized representative is capable of providing verbal confirmation of understanding the trial risks, benefits, and treatment alternatives associated with receiving immunosuppressive CAR-DC therapy, and provides written informed consent prior to participation in this clinical trial.

Exclusion Criteria（patients）:

1. Acute mechanical complications of infarction (e.g., ventricular septal rupture, acute mitral regurgitation).
2. Cardiac arrest.
3. Hypoxic-ischemic brain injury (cerebral injury with fixed and dilated pupils not attributable to medication).
4. Shock due to other causes (e.g., sepsis, hypovolemia).
5. Resuscitation duration >30 minutes.
6. Absence of spontaneous cardiac activity.
7. Persistent electrical instability.
8. Active bleeding or contraindications to heparin use.
9. Active autoimmune disease requiring immunosuppressive therapy.
10. History of malignancy.
11. Infection, including:

    * Active hepatitis B (HBV DNA >1000 copies/mL by PCR), hepatitis C, syphilis, or HIV infection at screening.
    * Uncontrolled systemic fungal, bacterial, viral, or other pathogen infections.
12. Pregnant women.
13. Contraindications to the investigational drug or study procedures.

Inclusion Criteria（donors）:

* Age ≥ 18 years and ≤ 75 years.
* Has provided written informed consent.
* Hematocrit >30%, lymphocyte count >0.5 × 10^9/L, platelet count >60 × 10^9/L.
* Pathogen screening results must be negative for HIV (antigen, core antibody, and RNA), HBV (surface antigen and core antibody), HCV, syphilis, CMV, and EBV.

Exclusion Criteria（donors）:

* Active infection requiring treatment.
* History of malignancy.
* Active autoimmune disease requiring immunosuppressive therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with Dose-limiting toxicity (DLT) | in 14 days after injection
  The proportion of participants with DLT as assessed by CTCAE v5.0
Incidence of treatment-emergent adverse events (TEAEs) | in 14 days after injection
  Incidence of iCDC treatment-emergent adverse events

SECONDARY OUTCOMES:
All-cause mortality | 30 days after injection
  All-cause mortality at 30 days after iCDC treatment
Systolic blood pressure | 24 hours、48 hours、72 hours、7 days after injection
  Systolic blood pressure (mmHg) measured using a calibrated sphygmomanometer under standardized conditions.
Diastolic blood pressure | 24 hours、48 hours、72 hours、7 days after injection
  Diastolic blood pressure (mmHg) measured using a calibrated sphygmomanometer under standardized conditions.
Mean arterial pressure | 24 hours、48 hours、72 hours、7 days after injection
  The mean arterial pressure (MAP) is calculated using the following formula:
  MAP=DBP+1/3(SBP-DBP)；DBP : Diastolic blood pressure，SBP ：Systolic blood pressure
Time to hemodynamic stability | From the end of the iCDC infusion to achievement of hemodynamic stability, assessed continuously until ICU discharge (up to 30 days).
  Sustained (> 60 min) systolic blood pressure >90 mmHg without requirement for catecholamines and without signs of peripheral endorgan hypoperfusion
Dose of vasopressors | 24 hours、48 hours、72 hours、7 days after injection
  Dose of vasopressors administered to the participant.
Duration of vasopressor use | From enrollment to hospital discharge (up to 30 days).
  Duration of vasopressor therapy in days treated with vasopressor between enrollment and hospital discharge. A day treated with vasopressor is any day during the hospital period where the patient received a vasopressor.
Dose of inotropic drugs | 24 hours、48 hours、72 hours、7 days after injection
  Dose of inotropic drugs administered to the participant.
Duration of inotropic drugs use | From enrollment to hospital discharge (up to 30 days).
  Duration of inotropic drugs therapy in days treated with inotropic drugs between enrollment and hospital discharge. A day treated with inotropic drugs is any day during the hospital period where the patient received inotropic drugs
Serum lactate level | The measurement frequency is once every 8 hours for a duration of 48 hours.
  Lactate is assessed via arterial blood gas analysis.
Change in B-type natriuretic peptide (BNP) level from baseline | 7 days，14 days，30 days after injection.
  Change in serum B-type natriuretic peptide concentration compared with baseline.
Change in C-reactive protein (CRP) level from baseline | 24 hours, 72 hours, 7 days，14 days after injection.
  Change in serum C-reactive protein concentration compared with baseline.
Change in serum creatinine level from baseline | 24 hours, 72 hours, 7 days，14 days after injection.
  Change in serum creatinine concentration compared with baseline.
Change in ALT (Alanine Aminotransferase) level from baseline | 24 hours, 72 hours, 7 days，14 days after injection.
  Change in serum ALT concentration compared with baseline.
Change in AST (Aspartate Aminotransferase) level from baseline | 24 hours, 72 hours, 7 days，14 days after injection.
  Change in serum AST concentration compared with baseline.
Change in Interleukin-6 (IL-6) levels from baseline | 24 hours, 72 hours, 7 days，14 days after injection.
  Change in serum Interleukin-6 (IL-6) levels compared with baseline.
Need for mechanical ventilation | From the end of the drug infusion until ICU discharge (up to 30 days).
  Need for mechanical ventilation is defined as requiring invasive or non-invasive positive pressure ventilation for at least 1 hour due to respiratory failure.
Duration of mechanical ventilation | From the initiation of mechanical ventilation until ICU discharge (up to 30 days).
  Duration of mechanical ventilation is defined as the total number of hours from the initiation of invasive or non-invasive ventilation until the last successful extubation
Requirement for left ventricular assist device implantation | From the end of iCDC infusion through study completion (up to 30 days).
  Requirement for left ventricular assist device implantation is defined as the need for implantation of a left ventricular assist device as bridge-to-transplant or destination therapy in patients with cardiogenic shock or end-stage heart failure who fail to maintain adequate end-organ perfusion despite optimized medical therapy.
Duration of left ventricular assist device use | From left ventricular assist device implantation through study completion (up to 30 days).
  Duration of left ventricular assist device use is defined as the total time from completion of device implantation until device removal, patient death, or the study cutoff date, whichever occurs first.
Simplified Acute Physiology Score II | Daily from ICU admission through ICU discharge (up to 30 days).
  The Simplified Acute Physiology Score II (SAPS II) is a validated severity-of-disease scoring system used to assess the physiological status of critically ill patients. The score ranges from 0 to 163, with higher scores indicating greater disease severity and a worse prognosis. SAPS II will be calculated based on the worst physiological values recorded during each 24-hour period.
time to recovery from cardiogenic shock | From the end of iCDC infusion to recovery from cardiogenic shock, assessed continuously until ICU discharge (up to 30 days).
  Time to recovery from cardiogenic shock is defined as the duration from the end of the single study drug infusion to the achievement of predefined criteria for hemodynamic stability and improvement in end-organ perfusion.
length of stay at the intensive care unit | From ICU admission until ICU discharge (up to 30 days).
  Length of stay in the ICU is defined as the total time from ICU admission until ICU discharge.
Length of hospital stay; | From hospital admission until hospital discharge or death (up to 30 days).
  Total hospital length of stay is defined as the total calendar days from patient admission registration until final discharge or death, whichever occurs first.
Left ventricular ejection fraction (LVEF) | 1 month after injection
  The difference of LVEF from baseline. LVEF will be assessed by echo.
SCAI Shock Classification | 3 days、7 days、14 days after injection
  The SCAI shock classification is a standardized, five-stage system (from A to E) used to categorize the severity of cardiogenic shock based on clinical, hemodynamic, and biomarker criteria.
assessment of heart failure symptom | 1 month after injection
  The difference of heart failure symptom, which will be assessed by NYHA grading and KCCQ score.
Incidence of major adverse cardiovascular events (MACE) | 1 month after injection
  Incidence of Cardiac death, readmission due to heart failure.
incidence of adverse events | From the end of the drug infusion through study completion，up to 30 days.
  Incidence of adverse events of heart, nerve system, mental system, digestive system and immune system.

CONTACTS AND LOCATIONS:
Overall Officials: Xinyang Hu, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No